CLINICAL TRIAL: NCT07237984
Title: Colorectal OmiCs and Oncofetal Chondroitin Sulfate-modified Proteoglycans in Screening and Colorectal Cancer Diagnostic Pathway
Brief Title: Colorectal Omics and ofCS Proteoglycans (COCO) in Screening and a Diagnostic Pathway
Acronym: COCO-S
Status: Not yet recruiting | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: COCO-S
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer; Colorectal Adenoma; Inflammatory Bowel Disease (IBD)
Keywords: Biomarker; Colorectal Cancer; Glycoproteins; Proteomics
MeSH Terms: conditions — Colorectal Neoplasms; Inflammatory Bowel Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood including plasma and serum, and stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Coloretcal Screening Patients: In the Danish national colorectal cancer screening programme a full colonoscopy is recommended within 14 days colon after a positive (Faecal Immunochemical Test, FIT) test, defined as >100 µg Hgb/L (20 µg Hgb/g feces).
  Patients referred to the study sites will be offered a single blood sample before bowel preparation for the colonoscopy.
  Interventions: Diagnostic Test: Blood sampling
- Colorectal Cancer Pathway Patients: In Denmark, patients with symptoms aligning with a suspicion of colorectal cancer are by law to be offered a full colonoscopy within 14 days.
  Patients referred to the study sites will be offered a single blood sample and a Faecal Immunochemical Test (FIT) before bowel preparation for the colonoscopy.
  Interventions: Diagnostic Test: Blood sampling; Diagnostic Test: Stool samplong

INTERVENTIONS:
Diagnostic Test: Blood sampling — Analyses of ofCS proteoglycans, proteomics (proteins), metabolomics (metabolits) and other biomarkers.
Diagnostic Test: Stool samplong — Fecal immunochemical test (FIT), feces sampled by the participant
  Groups: Colorectal Cancer Pathway Patients

SUMMARY:
Colorectal Cancer (CRC), or bowel cancer, is a serious disease that affects many people globally. The earlier CRC is diagnosed, the better the patient outcomes.

The problem with the current diagnostic methods is that they lead to many unnecessary endoscopies (colonoscopies). In Denmark alone, over 30,000 patients every year undergo a colonoscopy without having a serious disease. This puts a major strain on both patients and the healthcare system.

This research project aims to solve that problem. COCO-S is investigating oncofoetal chondroitin sulphate-modified proteoglycans (ofCS) to see if ofCS can be used as a novel, unique cancer marker found in the blood.

ofCS are special molecules that reappear in most tumour tissues. A method has been developed to detect ofCSs in a simple blood sample.

Initial findings from an ongoing study are highly promising. A test using five different ofCS markers has shown very high accuracy in detecting CRC: it correctly identifies 86% of cancer cases (sensitivity) and correctly gives a "negative" result in 97% of cases without cancer (specificity).

The results also suggest that high ofCS levels might help clinicians detect adenomas (polyps), which are early precursors to cancer.

Combining the analysis of ofCS in the blood with the existing stool test (FIT) and other promising blood markers can significantly improve patient selection for a colonoscopy.

This project will collect blood samples from patients scheduled for a colonoscopy. The blood will be analysed for ofCS and other substances to determine the combined predictive value for patients who truly require the procedure.

The findings from this project could revolutionize CRC diagnosis. By more accurately identifying patients who need a colonoscopy, the number of unnecessary, invasive procedures can be reduced while maintaining patient safety and ensuring cancer is found in time.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is a significant global health burden. Early detection improves outcomes, but current diagnostic pathways lead to many unnecessary colonoscopies. In Denmark, over 30,000 colonoscopies are performed annually on patients without any pathology, burdening both healthcare resources and patients.

This project aims to address this unmet clinical need by investigating the potential of oncofoetal chondroitin sulphate-modified proteoglycans (ofCS) as a novel, tumour-specific biomarker for improved patient allocation to colonoscopy. OfCS are unique molecules that re-emerge in most cancer tissues and can be detected in blood plasma using a proprietary method developed.

Preliminary findings from an ongoing study in CRC patients are highly encouraging. A panel of five ofCS biomarkers has shown high accuracy in detecting CRC, with a cumulative AUC of 0.96, a sensitivity of 86%, and a specificity of 97%. Importantly, these results also suggest that elevated ofCS levels may help detect adenomas, an early precursor to CRC.

Incorporating ofCS analysis into existing diagnostic frameworks, such as the faecal immunochemical test (FIT), will significantly improve the accuracy of patient selection for colonoscopy.

The study assesses whether supplementing the FIT with ofCS analysis and other biomarkers from proteomics and metabolomics can yield a significantly higher AUC of the receiver operating characteristic (ROC) in both the screening and the 'cancer patient pathway'.

This prospective cohort study includes patients undergoing a colonoscopy. Participants blood will be analysed for ofCS, and proteomics and metabolomics biomarkers, to determine their combined predictive value.

The findings from this project could revolutionise CRC diagnosis by creating a tailor-made pathway. By more accurately identifying patients who need a colonoscopy, invasive procedures can be reduced while maintaining patient safety and cancer detection rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned to undergo a colonoscopy either as part of the colorectal cancer screening programme due to a positive FIT or within a 'cancer patient pathway' for CRC at one of the study sites.
* Able to speak Danish, English, or other languages with sufficient interpretation provided by relatives.
* Able to give informed consent

Exclusion Criteria:

* Patients previously included in the study
* Patients known to be pregnant (pregnancy test not required)
* Non-resident in Denmark.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People living within the Capital Region of Denmark referred to a screening or colorectal cancer diagnostic pathway colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Colorectal cancer | 30 days
  The value of ofCS proteoglycans in blood plasma as a diagnostic test of finding colorectal cancer at colonoscopy
Colorectal adenoma | 30 days
  The value of ofCS proteoglycans in blood plasma as a diagnostic test of detecting adenomas at colonoscopy

SECONDARY OUTCOMES:
Inflammatory bowel disease | 30 days
  The value of ofCS proteoglycans in blood plasma as a diagnostic test of finding inflammatory bowel disease at colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Claus Anders Bertelsen, PhD MD, Study Chair — Copenhagen University Hospital - North Zealand
Locations (2):
- Denmark (2):
  - Copenhagen University Hospital - North Zealand, Hillerød
  - Copenhagen University Hospital - Amager-Hvidovre, Hvidovre

IPD SHARING:
Plan to Share IPD: Yes